CLINICAL TRIAL: NCT03575078
Title: PHASE 1 DOSE ESCALATION TRIAL OF β-LAPACHONE (ARQ761) IN COMBINATION WITH PARP INHIBITOR, OLAPARIB, FOR REFRACTORY, ADVANCED SOLID TUMORS
Brief Title: ARQ761 + PARP Inhibitor in Refractory Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Project Never Initiated - no human subjects were enrolled and no data regarding humans was collected or studied
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 052018-073
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: Phase 1 Dose Escalation
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Maximum tolerated dose of ARQ761 in combination with Olaparib. (Experimental): ARQ761: weekly infusion. Olaparib Dose 1 D-7 administered orally twice daily
  Interventions: Drug: ARQ761, Olaparib

INTERVENTIONS:
Drug: ARQ761, Olaparib — ARQ761: weekly infusion. Olaparib Dose 1 D-7 administered orally twice daily

SUMMARY:
Open Label, dose escalation in a 3+3 study design to establish the RP2D of the combination of ARQ761 and a PARP inhibitor, Olaparib

DETAILED DESCRIPTION:
Open Label, dose escalation in a 3+3 study design to establish the RP2D of the combination of ARQ761 and a PARP inhibitor, Olaparib. This is an exploratory Phase 1 trial evaluating the safety and tolerability of the combination of ARQ761 and Olaparib.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Patients with histologically or cytologically confirmed locally advanced or metastatic solid tumors that have received standard of care for their disease and for which no other approved therapy is available or if patient has declined other approved therapies.
* Age ≥ 18 years.
* Performance status ECOG 0-1.
* Measurable disease as per RECIST criteria 1.1.
* Access to archival tissue (available unstained slides of tumor tissue).
* Central venous access, such as a Portacath or Hickman Line.
* Adequate organ and marrow function measured within 14 days prior to administration.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
* Has not undergone a hysterectomy or bilateral oophorectomy; or Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and willing to sign a written informed consent. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
* Patients must have a life expectancy ≥ 16 weeks.
* At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.
* Postmenopausal is defined as:

  1. Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
  2. Luteinizing Hormone (LH) and Follicle Stimulating Hormone (FSH) levels in the post-menopausal range for women under 50
  3. Radiation-induced oophorectomy with last menses >1 year ago
  4. Chemotherapy-induced menopause with >1 year interval since last menses
  5. Surgical sterilization (bilateral oophorectomy or hysterectomy)

Exclusion Criteria:

* Those whose adverse events from prior therapies have not recovered to ≤ grade 1 except alopecia.
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment.
* Concurrent therapy: No other concurrent anticancer or investigational therapy permitted except as noted above.
* Subjects with known, untreated and/or symptomatic brain metastases: Subjects with known, treated brain metastases must be stable with no symptoms for four weeks after completion of treatment, with image documentation required, and must either be off steroids or on a stable dose of steroids for at least two weeks prior to protocol enrollment.
* Subjects with known leptomeningeal metastases are excluded, even if adequately treated.
* Patients with spinal cord compression are excluded unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
* Subjects without known brain metastases do not require radiologic imaging prior to enrollment.
* Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, significant pulmonary disease (shortness of breath at rest or mild exertion), uncontrolled infection or psychiatric illness/social situations that would limit compliance with study requirements.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agent(s) or other agents used in study.
* Pregnant or nursing subjects due to the potential for either congenital abnormalities or harming infants who are being nursed, respectively.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca, ArQule staff and/or staff at the study site).
* Previous enrollment in the present study.
* Participation in another clinical study with an investigational product during the last 4 weeks.
* Any previous treatment with PARP inhibitor, including olaparib.
* Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome.
* Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
* Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Breast feeding women.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients with a known hypersensitivity to ARQ761.
* Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable per 3.1.8).
* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years.
* Patients with a history of localized triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of ARQ761 in combination with Olaparib. | Day 1-28
  If a dose limiting toxicity (DLT) is observed in 1 out of 3 patients at a given dose level, up to 3 additional patients will be enrolled and treated at that dose level.

SECONDARY OUTCOMES:
Dose limiting toxicities | 4 weeks
  DLT will be defined by the occurrence of any of the following toxicities possibly or probably related to treatment, during cycle 1 only:
  Grade 3 or 4 hemolysis or hemolytic anemia, except: Transfusion for hemolysis or hemolytic anemia will be considered a DLT only if Hgb < 8.0 g/dL (Grade 3 anemia) (b) Any drug related grade 3 or grade 4 non-hematological toxicity, except alopecia, nausea, diarrhea and vomiting in the absence of optimal anti-diarrheal and/or anti-nausea medications (c)Grade 4 neutropenia lasting more than 7 days. (d) Platelets <50,000/µl for longer than 7 days or any platelet count <25,000/µl. (e) Grade 3 or 4 hyperbilirubinemia that does not recover to Grade 1 within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Beg, Principal Investigator — UTexas Southwestern